CLINICAL TRIAL: NCT00467324
Title: The Advance Trial. Tongue Advancement for Obstructive Sleep Apnea: An Evaluation of the Aspire Medical Advance System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aspire Medical (Industry)
Responsible Party: Jafar Shenasa, Director, Clinical and Regulatory Affairs, Aspire Medical, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS 002
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apnea; surgery; tongue
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Aspire Medical Advance System — The treatment includes a device that is surgically implanted in the tongue and lower jaw. The purpose of the implant is to prevent obstruction of the upper airway thereby improving breathing during sleep.

SUMMARY:
The objective of the study is to assess the effectiveness of the Aspire Medical Advance System in obstructive sleep apnea by demonstrating a statistically significant mean reduction in the apnea-hypopnea index (AHI) from baseline to 6 months, measured by polysomnography (PSG).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a major health problem in the United States and can result in excessive daytime sleepiness and cardiovascular problems. The primary treatment for OSA today is continuous positive airway pressure (CPAP). Many patients however are unable to tolerate sleeping with a CPAP machine. Surgery is one of the main treatment options available today to these CPAP-intolerant patients. However, current methods of sleep surgery are painful, morbid, and/or lack decent effectiveness.

This trial will measure the effectiveness of the Advance System, an implantable medical device to treat OSA. In the trial, patients who meet the study entry criteria receive a baseline sleep study (PSG). The Advance System is then implanted and 6 months after implantation, another PSG is performed. The trial will compare the baseline and the 6 month apnea-hypopnea indices

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed or screened with moderate to severe sleep apnea who have an AHI of between 15 and 60
* Age between 18 and 65
* Body mass index (BMI) </= 32
* Patient has been offered CPAP and has refused or failed to continue CPAP treatment
* Identified evidence of airway collapse at the base of the tongue
* Signed informed consent

Exclusion Criteria:

* Prior OSA surgery except tonsillectomy, adenoidectomy, and nasal surgery
* Enlarged tonsils (3+ and 4+)
* Anatomy unable to accommodate the implant
* Severe mandibular deficiency/retrognathia
* Significant rhinitis/nasal obstruction
* Unable and/or not willing to comply with treatment follow-up requirements
* Pregnancy (female subjects of childbearing age mus have a negative pregnancy test prior to enrollment and should maintain adequate contraception during the study) or breastfeeding
* Active systemic infection
* Allergy to latex or any medication used during implantation
* Previous history of neck or upper respiratory tract cancer
* History of radiation therapy to neck or upper respiratory tract
* Dysphagia
* History of major cardiovascular disorders including MI, angina, uncontrolled hypertension, and CHF
* Major pulmonary disorders including COPD and uncontrolled asthma
* Patient is suffering from untreated/inadequately treated major depression, as determined by history
* History of falling asleep driving or motor vehicle accident secondary to excessive sleepiness
* Anesthesia risk group ASA Class IV or V
* Other medical, social or psychological problems that, in the opinion of the investigator, could complicate the procedure and/or recovery from this treatment or could complicate the procedures and evaluations pre- and post-treatment
* Enrollment in another pharmacological or medical device study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea index measured with polysomnography 6 months after implantation of the Advance System | 6 months

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) measured at 6 months post-implantation | 6 months
Functional Outcomes of Sleep Questionnaire (FOSQ) measured at 6 months post-implantation | 6 months
Safety: assessment of all device-related and procedure related adverse events and their seriousness | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tucker Woodson, MD, Principal Investigator — Department of OTO-HNS Medical College of Wisconsin
Locations (4):
- United States (4):
  - Northside Hospital/Advanced Ear Nose & Throat Associates PC, Atlanta, Georgia
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Sponsor's web site; has basic product & patient information — http://www.aspiremedical.com